CLINICAL TRIAL: NCT00425633
Title: A Study To Evaluate The Effect Of Homeopathic Concentrations Of Potassium Dichromate On Tracheal Secretions In Critically Ill Patients.
Brief Title: Efficacy Study of Homeopathic Potassium Dichromate to Treat Tracheal Secretions in Critically Ill Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sharon Yamashita Pharm.D., Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 418-2006
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Ventilator Adverse Event
Keywords: Homeopathic; Potassium; Dichromate; Kalium; Bichromicum; Mechanical; Ventilation; Secretions
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Homeopathic Potassium Dichromate — 5 pellets under tongue q12h until extubation

SUMMARY:
The purpose of this study is to find out whether homeopathic potassium dichromate will decrease the time on the breathing machine and the amount of phlegm that you produce in your lungs. In addition, this study will look at whether participants spend less time in a critical care unit and if the chances of being placed back on a breathing machine can be lessened.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation is associated with greater mortality, increased need for tracheostomy, prolonged length of critical care stay and higher costs. Risk factors identifying patients at greater risk of unsuccessful extubation include cough strength, endotracheal secretions and neurological status. These factors are synergistic and patients exhibiting two of the above determinants have an extubation failure rate of 81%. The risk is 100% if all three are present as compared to 3% in a patient with no risk factors. Several strategies including administration of mucolytics, anti-cholinergics and corticosteroids have met with limited success or excessive toxicity. Thus, methods to improve the quality and quantity of secretions could be associated with decreased extubation failure and greater overall outcomes.

The most recent study was a randomized, double blind, placebo controlled trial of 50 critically ill ventilated patients with a previous history of COPD and tobacco use by Frass et al. Five C30 pellets of potassium dichromate or placebo were administered twice daily until extubation and it was found that those receiving the homeopathic formulation had statistically significant (p<0.0001) tracheal secretion reductions, earlier extubation times and shorter lengths of stay in critical care as compared to their placebo counterparts.

Use of homeopathy in the critically ill would convey a number of advantages including lack of adverse effects or drug interactions, due to the dilute nature of the solutions, and be a cost effective adjunct to conventional therapy. In the previous trial of potassium dichromate in critical care patients, only patients with previous tobacco use and history of COPD were included. It is unknown whether those results could be extrapolated to the general critical care population.

Therefore, this study will look at the safety and efficacy of homeopathic potassium dichromate (Kalium Bichromicum)vs placebo. A dosing schedule of five pellets every 12 hours will be utilized; this regimen was chosen based on previous evidence showing efficacy at this dose. Dosing will continue until the patient is extubated or chooses to withdraw from the study. Data collected will include baseline demographic data, quantity of sputum production (at baseline and per day), number of times suctioning required per day, duration of mechanical ventilation, rate of reintubation within 7 days following extubation, critical care length of stay, PaO2/ FiO2 ratios, PaCO2 twice daily, and number of therapeutic bronchoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18yrs and older
* Situated in the Critical Care areas of Sunnybrook Health Sciences Centre including the Critical Care Unit, Cardiovascular Surgery Intensive Care Unit, Ross Tilley Burn Centre and B5/D4 intensive care units.
* They will have been weaned from mechanical ventilation (eg: extubated, face mask or tracheostomy mask, minimal pressure support or CPAP, FiO2 <0.3) but are unable to be transferred out of the unit due to excessive and/or persistent secretions for at least 48 hours.
* Persistent secretions will be defined as suctioning of greater than every 2 hours or a score of greater than 20-24 "MP" per day. (In the Critical Care areas, each time a patient is suctioned, secretions are quantified on a scale of 1-3, with "MP" being mucopurulent in nature).

Exclusion Criteria:

* Those with evidence of untreated respiratory infections or infections treated for less than 48 hours.
* Those patients on high dose steroids as defined by greater than:Fluticasone 125ug inhaler- four puffs twice daily and/or Prednisone 20mg daily orally
* Patients with multiple drug and/or environmental allergies
* Those patients who fail to give informed written consent.
* Those patients currently enrolled in another clinical trial or who have been approached for participation in a trial during the last 30 days.
* Previous enrollment in this study
* Pregnancy- all women of child bearing age will be administered a pregnancy test before inclusion into the study to verify their status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of potassium dichromate on the quantity of tracheal secretions. | until extubation

SECONDARY OUTCOMES:
To evaluate the efficacy of homeopathic potassium dichromate on duration of mechanical ventilation, required suctioning per day, re-intubation rate, length of ICU admission and number of therapeutic bronchoscopies required. | until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Yamashita, PharmD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Frass M, Dielacher C, Linkesch M, Endler C, Muchitsch I, Schuster E, Kaye A. Influence of potassium dichromate on tracheal secretions in critically ill patients. Chest. 2005 Mar;127(3):936-41. doi: 10.1378/chest.127.3.936. PMID 15764779